CLINICAL TRIAL: NCT05111457
Title: Injury Prevalence and Risk Factors in Swedish Padel Recreational and Competition Players
Brief Title: Injuries in Swedish Padel
Status: Completed | Type: Observational
Sponsor: Sofia Ryman Augustsson (Other)
Responsible Party: Sponsor-Investigator, Sofia Ryman Augustsson, Associate Professor, Linnaeus University
Organization: Linnaeus University (Other)
Other Study IDs: 2021-03382
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Injury;Sports
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project is to investigate the injury panorama of acute and overuse injuries in women and men who regularly participate padel. The intention is to provide insights on injury prevalence, injury location, injury consequences, gender differences and risk factors .

This study will be conducted as a retrospective cohort study where the participants consist of female and male padle players, both at the recreational and competition level, with at least 6 months' experience in the sport. The information from this project can be valuable in the work of identifying risk factors for padle injuries and injury prevention strategies.

DETAILED DESCRIPTION:
Study design and participants This study will be conducted as an observational study using a retrospective survey. The participants will consist of padle players at both recreational and competitive level. An estimated 300 players will participate (~ 50% women). Recruitment will take place through inquiries via padle associations, social media and information flyers posted on padle courts around the Stockholm and Kalmar region. The survey will be aimed at all regularly active women and men padle players, aged 18-65, with at least 6 months' experience in the sport. Players with <1 hour of padle training per week will be excluded.

Procedure During the autumn of 2021, data collection will start for the retrospective part and then continue for about 3 months. Injury registration will be carried out using a web-designed registration form (SurveyMonkey®). The survey is designed with a previously developed form for acute injuries and with the help of the online survey OSTRC Overuse Injury Questionnaire for injuries of an overuse nature. The participant will register any musculoskeletal injury and complaints that have occurred during the last 6 months. The players will also provide information about age, gender, number of training hours per week and experience of padle and other training routines.

Injury definition The injuries will be classified as either traumatic, i.e., the player could define a specific sudden onset of pain with a defined trauma included, or as due to overuse. The severity of the injury will be graded by the time of absence from training and match participation. The injuries will be divided into three categories. ''Minor'' is defined as an injury leading to an absence from training/matches of no more than 1 week. Injury leading to an absence of 2-4 weeks is defined as ''moderate''. ''Major'' is defined as an injury leading to an absence of more than 4 weeks.

Measurements The OSTRC survey was developed in Norway and has been translated and validated into Swedish. The sensitivity of this survey is assumed to be much greater than traditional questionnaires about injuries in sports and enables more overload injuries to be identified. In addition, the survey registers the extent of injury prevention strategies as well as training frequency, intensity, amount and type of training. The body regions that will be registered are neck, shoulder, elbow, hand/wrist, thoracic spine, lumbar spine, hip, thighs, knees and lower legs and foot/ankle. Participants will also estimate the severity of the problems on ordinal scale ranging from 0-4, where "0" is referring to no problem, for each body region. The acute injuries will be registered using previously developed forms for acute injuries.

Statistics Statistics will be calculated using SPSS®25.0 (IBM SPSS Statistics, New York, USA). Descriptive statistics (mean ± SD and range) will be calculated for each variable. To compare means between the groups (women and men, age groups, recreational versus competitive players), independent student T-tests will be used. Fisher's exact test will be used to compare different injury location between groups. Pearson's correlation coefficient will be used to assess associations between variables.To calculate if data is normally distributed, in the retrospective part, a Shapiro-Wilks test of normality will be performed. The level of significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Regularly active women and men padle players
* Aged 18-65
* At least 6 months' experience in padel.

Exclusion Criteria:

* Players with <1 hour of padle training per week.
* Players with less then 6 months' experience of padle training.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will consist of padle players at both recreational and competitive level. An estimated 300 players will be invited to participate (~ 50% women). Recruitment will take place through inquiries via padle associations, social media and information flyers posted on padle courts around the Stockholm and Kalmar region.
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Injuries occured during padel; training and/or match | Injuries during the last 6 month
  Prevalence (number) of acute and overuse injuries
Body region injured | Last 6 month
  Description of body region injured and prevalence; number of injuries at one site/of total number of injuries

SECONDARY OUTCOMES:
Type of injury | Last 6 month
  Number of different types of injury, prevalence; number of a specific type of injury/of total number of injuries
Injury occurence in relation to different enviroment | Last 6 month
  Prevalence (number) of acute and overuse injuries in relation to different enviroment
Injury occurence in relation to different padel rackets | Last 6 month
  Prevalence (number) of acute and overuse injuries in relation to different rackets
Sex difference in injury occurence | Last 6 month
  Prevalence (number) of acute and overuse injuries in men versus women

CONTACTS AND LOCATIONS:
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden